CLINICAL TRIAL: NCT01719029
Title: Role of Macronutrient Diet Composition on Maternal and Infant Metabolic Outcomes in Gestational Diabetes
Brief Title: Role of Macronutrient Diet Composition and Infant Metabolic Outcomes in Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07-0283
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Gestational Diabetes Mellitus
Keywords: continuous glucose monitoring; gestational diabetes; diet therapy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Diet (Experimental): Low carbohydrate/higher fat diet: 40% carbohydrate, 45% fat, 15% protein
  Interventions: Other: High Carbohydrate/Low fat diet
- Complex Carbohydrate Diet (Experimental): High complex carbohydrate/lower fat diet: 60% complex carbohydrate, 25% fat, 15% protein
  Interventions: Other: Low-Carbohydrate/Higher Fat Diet

INTERVENTIONS:
Other: Low-Carbohydrate/Higher Fat Diet
  Arms: Complex Carbohydrate Diet
Other: High Carbohydrate/Low fat diet
  Arms: Conventional Diet

SUMMARY:
A better understanding of the optimal diet for women with gestational diabetes is fundamental to the management of this rapidly growing problem in pregnancy. Careful comparison studies of the current low- carbohydrate, higher-fat diet versus a diet higher in complex carbohydrate but lower in fat is critical in order to determine which diet results in a more favorable maternal 24-hour glucose, lipid, and inflammatory profile, all of which directly effect optimal fetal growth and may influence the future health of the offspring.

DETAILED DESCRIPTION:
Despite the doubling in the prevalence of gestational diabetes mellitus (GDM) over the last 10 years, dietary management guidelines remain ambiguous due to the paucity of randomized controlled trials. New diagnostic criteria recently developed for the diagnosis of GDM are expected to increase the prevalence to 10-15% of all pregnant women. There is growing recognition that GDM has long-term implications on maternal risk for diabetes and that the intrauterine GDM environment is an independent risk factor for childhood obesity and impaired glucose tolerance. Yet, how diet can be used to modify fetal fuel and attenuate this risk remains unknown in humans. Fundamental to the management of GDM is dietary intervention, yet the historic practice of advising a low-carbohydrate (CHO), higher-fat diet has not been sufficiently tested. Both animal and non-human primate data support a fetal programming influence that maternal high-fat diets may promote insulin resistance, glucose intolerance, and hepatic steatosis in the offspring. Recent human data suggest that high maternal triglycerides (TG) and free fatty acids (FFA), variables sensitive to dietary manipulation, are independent risk factors for fetal macrosomia and adiposity. As a result, consensus groups have abandoned any specific diet recommendations for women with GDM. Despite the pivotal role of diet therapy in the treatment of GDM, no randomized trials have directly compared glycemic and lipoprotein profiles of the conventional higher-fat diet with any other diet. To address this critical need, the aims of this randomized cross-over trial are to study the effects of a high complex carbohydrate/low-fat diet (HC/LF; 60% CHO, 25% fat, 15% protein) compared to the usual care, low-CHO/higher fat diet (LC/HF; 40% CHO, 45% fat, and 15% protein) in GDM women on: 1) 72-hour glycemic profiles using a continuous glucose monitoring system within subjects; 2) postprandial lipemia by measuring serial plasma TG and FFA over a 5-hour, post-breakfast meal period within subjects; and 3) maternal lipoproteins, inflammatory profiles, and in-vitro adipose tissue lipolysis after 6-8 weeks of diet therapy between subjects. We will also measure neonatal adiposity by air displacement plethysmography and newborn markers of lipid peroxidation, inflammation, and dietary fat intake in the babies born to mothers with GDM. This pilot study will directly test which GDM diet is most effective in limiting maternal hyperglycemia and hyperlipidemia in a randomized controlled fashion, potentially optimizing fetal substrate availability and fetal growth. Our goal is to determine which diet intervention might favorably impact a cycle that could otherwise perpetuate future diabetes, obesity, and CVD in both mother and offspring.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria. Potential participants will be ≥ 0-36 years old, which includes the offspring of the pregnant mothers with GDM. Pregnant women will be between the ages of 18-40 years and will have a BMI of 26 - 35 kg/m2 at the time of diagnosis, a singleton pregnancy, and will not be taking medication for their GDM on entrance to the study. Subjects will have been diagnosed with GDM according to the criteria established by the ADA and the ACOG (19;35;53), specifically, they will meet the following criteria:

* A 50-gram Glucola in which the one hour reading is >200 mg/dL and the FBG is >95 mg/dL
* Two abnormal values on a 100-gram 3 hour glucose tolerance test based on the Coustan and Carpenter criteria as adopted by the ADA and Fourth International Workshop on Gestational Diabetes (76;77):

  * Fasting > or = to 95 mg/dL but <126 mg/dL
  * 1 hr >/= 180 mg/dL
  * 2 hr >/= 155 mg/dL
  * 3 hr >/=140 mg/dL

Exclusion Criteria:Those women with overt diabetes and those suspected of having preexisting diabetes by any of the following criteria will be excluded, including:

* Fasting glucose >110 mg/dL, due to the high likelihood of rapidly failing diet and requiring medical treatment (35).
* Random glucose > 200 mg/dL
* Glycosylated hemoglobin A1C > 6.5
* Non-English speaking patient
* Fasting TG > 400 mg/dL

Women who smoke will be excluded since this is the leading cause of low birth weight. In addition, women with other risk factors for placental insufficiency, including hypertension requiring beta-blocker treatment, renal disease, thrombophilias, preeclampsia, steroid use, history of pancreatitis or infectious disease such as hepatitis, or intrauterine growth restriction will be excluded.

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2007-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Glucose area-under-the-curve | During 3 days of each diet treatment
  The average glucose area-under-the-curve over 3 days, calculated using 24-hour continuous glucose monitoring

SECONDARY OUTCOMES:
Infant Adiposity | 2 weeks after birth
  Infant adiposity measured using Pea Pod

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Derived] Hernandez TL, Van Pelt RE, Anderson MA, Reece MS, Reynolds RM, de la Houssaye BA, Heerwagen M, Donahoo WT, Daniels LJ, Chartier-Logan C, Janssen RC, Friedman JE, Barbour LA. Women With Gestational Diabetes Mellitus Randomized to a Higher-Complex Carbohydrate/Low-Fat Diet Manifest Lower Adipose Tissue Insulin Resistance, Inflammation, Glucose, and Free Fatty Acids: A Pilot Study. Diabetes Care. 2016 Jan;39(1):39-42. doi: 10.2337/dc15-0515. Epub 2015 Jul 29. PMID 26223240